CLINICAL TRIAL: NCT06965777
Title: The Space Changes Following Premature Loss of Lower First Primary Molars in the Primary Dentition Stage Using Digital Scanning A Prospective Split-mouth Clinical Study
Brief Title: Space Changes After Premature Loss of Lower First Primary Molars in Children Using Digital Scanning
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dania Yaser Rahhal, Principal Investigator, Cairo University
Other Study IDs: SL&AP-CU
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Premature Loss of Primary Molars; Space Maintenance; Dental Arch Development; Pediatric Tooth Extraction
Keywords: Tooth Loss; Dental Arch; Pediatric Dentistry; Primary Dentition
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Split-mouth Observational Cohort: Children aged 3 to 5.5 years with one mandibular first primary molar extracted due to poor prognosis. The study compares space and arch perimeter changes between the extraction side and the contralateral intact side within the same patient over a 6-month follow-up period using digital 3D models.

SUMMARY:
This prospective split-mouth clinical study aims to evaluate space changes in the mandibular dental arch following premature extraction of the lower first primary molar in children aged 3 to 5.5 years. Using digital 3D models, changes in the D space and mandibular arch perimeter will be measured at baseline and 6 months post-extraction. The goal is to determine whether space maintainers are necessary in the primary dentition stage.

DETAILED DESCRIPTION:
Premature loss of primary molars in children is a common result of caries or trauma, potentially affecting future occlusion and alignment. This study investigates the space changes that occur after unilateral premature extraction of the mandibular first primary molar before the eruption of the permanent first molar. Using a split-mouth design, the contralateral non-extracted side serves as the control. Digital impressions will be taken at baseline (day of extraction) and after 6 months. The primary outcome is the change in the D space, and the secondary outcome is the change in the mandibular arch perimeter, both measured using 3D digital software. The study aims to provide evidence for or against the routine use of space maintainers in similar clinical scenarios, potentially reducing unnecessary treatment and improving patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 5.5 years
* Mandibular first primary molar indicated for extraction due to extensive decay or hopeless prognosis
* Contralateral mandibular first primary molar must be intact and free of proximal caries
* No eruption of mandibular permanent first molar at the time of enrollment
* Presence of primary canines and second primary molars
* No space maintainers placed
* Parents/caregivers unable or unwilling to fabricate a space maintainer

Exclusion Criteria:

* Bilateral premature loss of mandibular first primary molars
* Contralateral mandibular molar has proximal caries or poor prognosis
* Children with good prognosis first primary molars (i.e., not needing extraction)
* Eruption of the mandibular permanent first molar
* Children who already have space maintainers
* Uncooperative behavior preventing study participation

Ages: 3 Years to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3 to 5.5 years attending the Pediatric Dentistry and Dental Public Health outpatient clinics at the Faculty of Dentistry, Cairo University, who require unilateral extraction of the mandibular first primary molar due to poor prognosis and meet the study's inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in D Space (Mandibular Arch) | Baseline (Day of Extraction) and 6 Months Post-Extraction
  The change in D space (distance between the mesial midpoint of the second primary molar and the distal midpoint of the primary canine) on the extraction side of the mandibular arch. Measured in millimeters using 3D digital models.

SECONDARY OUTCOMES:
Change in Mandibular Arch Perimeter | Baseline (Day of Extraction) and 6 Months Post-Extraction
  The change in the total arch perimeter of the mandibular arch measured using 3D digital models. The arch perimeter is calculated as the sum of linear segments across reference tooth landmarks. Measured in millimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPD). All data collected will remain confidential and used solely for the purposes of this research. Any results presented will be in aggregate form, without disclosing participant-level data.